CLINICAL TRIAL: NCT00682513
Title: Clinical, Genetic, and Cellular Consequences of Mutations in the NA,K-ATPase ATP1A3
Brief Title: Studies of the Variable Phenotypic Presentations of Rapid-Onset Dystonia Parkinsonism and Other Movement Disorders
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Allison Brashear, MD, MBA, Dean, Jacobs School of Medicine and Biomedical Sciences, State University of New York at Buffalo
Other Study IDs: 1688159; BG05-556 (Other: Wake Forest University School of Medicine); 1R01NS058949-01A1 (NIH); IRB00007686 (Other: Wake Forest University School of Medicine); 1704511 (Other: University of California, Davis IRB)
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2024-04

CONDITIONS: Dystonia; Parkinsonism
Keywords: dystonia; parkinsonism; rapid-onset dystonia-parkinsonism; RDP; Alternating Hemiplegia of Childhood; AHC
MeSH Terms: conditions — Dystonia; Parkinsonian Disorders; Dystonia 12; Alternating hemiplegia of childhood

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, tissue (saliva samples)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ATP1A3 Mutation: Those with RDP, AHC, unaffected carriers of ATP1A3 mutations, and non-carrying family members

SUMMARY:
The purposes of this study are to identify persons with rapid-onset dystonia-parkinsonism (RDP) or mutations of the RDP gene, document prevalence of the disease, and map its natural history.

DETAILED DESCRIPTION:
Rapid-onset dystonia-parkinsonism (RDP) is a rare, movement disorder with variable characteristics ranging from sudden onset (hours to days) of severe dystonic spasms to gradual onset of writer's cramp. RDP has elements of both dystonia and Parkinson's disease-two neurological diseases with motor and neuropsychological symptoms that hinder the quality of life. An internal trigger associated with extreme physiological stress has been reported prior to abrupt symptom onset of RDP.

This study, which is a continuation of an earlier study begun by Dr. Allison Brashear, aims to more clearly identify the characteristics associated with RDP and to explore whether mutations in the RDP gene are associated with atypical dystonias, Parkinson's disease, and other movement disorders.

The study involves in-person or remote (telemedicine) neurological assessments and blood samples for genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* clinical presentation consistent with ATP1A3 disease (RDP, AHC) or confirmed diagnosis of RDP or AHC

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Selection will take place predominantly via primary care clinics, i.e., physician referrals when patients present with a movement disorder suspicious for RDP.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2008-04; Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
RDP Severity | Visit 1 (baseline)
  History of symptom onset and duration will be obtained and current degree of severity assessed.

SECONDARY OUTCOMES:
Presence of neuropsychiatric disease | Will be assessed at Visits 1 (baseline) and 2 (24 months), approximately 2 years apart
  Psychiatric interview and cognitive assessment will be performed to examine presence or absence of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Brashear, MD, Principal Investigator — Dean, University at Buffalo Jacobs School of Medicine and Biomedical Sciences
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - University at Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cook JF, Hill DF, Snively BM, Boggs N, Suerken CK, Haq I, Stacy M, McCall WV, Ozelius LJ, Sweadner KJ, Brashear A. Cognitive impairment in rapid-onset dystonia-parkinsonism. Mov Disord. 2014 Mar;29(3):344-50. doi: 10.1002/mds.25790. Epub 2014 Jan 16. PMID 24436111
- [Derived] Brashear A, Mink JW, Hill DF, Boggs N, McCall WV, Stacy MA, Snively B, Light LS, Sweadner KJ, Ozelius LJ, Morrison L. ATP1A3 mutations in infants: a new rapid-onset dystonia-Parkinsonism phenotype characterized by motor delay and ataxia. Dev Med Child Neurol. 2012 Nov;54(11):1065-7. doi: 10.1111/j.1469-8749.2012.04421.x. Epub 2012 Aug 28. PMID 22924536
- See also: ATP1A3 diseases study website — http://www.atp1a3diseases.org/